CLINICAL TRIAL: NCT06225427
Title: Phase I Study of Gilteritinib for ALK Positive Non-Small Cell Lung Cancer
Brief Title: Gilteritinib for the Treatment of ALK NSCLC
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2023.047; NCI-2023-10639 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UMCC 2023.047 (Other: University of Michigan Comprehensive Cancer Center)
Record Dates: First submitted 2024-01-13; First posted 2024-01-26 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Lung Non-Small Cell Carcinoma; Stage IV Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Biopsy; Specimen Handling; gilteritinib; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (gilteritinib) (Experimental): Patients receive gilteritinib PO QD on days 1-21 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo echocardiography at screening and blood sample collection, CT scan and MRI at screening and on study. Additionally, patients may undergo a tumor biopsy pre-treatment and at end of treatment.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography; Drug: Gilteritinib; Procedure: Magnetic Resonance Imaging; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biopsy — Undergo tissue biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Procedure: Echocardiography — Undergo echocardiography
  Other Names: EC
Drug: Gilteritinib — Given PO
  Other Names: ASP-2215; ASP2215
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase I trial is studying the safety, side effects, and best dose of gilteritinib in treating patients with stage IV ALK positive non-small cell lung cancer (NSCLC) who have progressed on other treatments. While there are many approved targeted drugs for ALK NSCLC, resistance to these drugs frequently occur. Giltertinib is a drug that is already FDA approved for the treatment of a specific type of leukemia. However, studies using ALK positive lung cancer cells demonstrate activity of gilteritinib against these resistant cells. Therefore, in this clinical trial, the investigators plan to study the effect of giltertinib in patients with ALK NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Stage IV (American Joint Committee on Cancer [AJCC] 8th edition) non-small cell lung cancer with an oncogenic ALK fusion
* Histologies include adenocarcinoma, squamous cell carcinoma, adenosquamous adenocarcinoma, and NSCLC NOS (not otherwise specified)
* The presence of an oncogenic ALK fusion established from any Clinical Laboratory Improvement Act (CLIA) certified laboratory
* The patient must belong to one of the following treatment cohorts.

  * Cohort 1: Prior 1st generation ALK tyrosine kinase inhibitor (TKI) (crizotinib) and/or prior 2nd generation TKI (ceritinib, brigatinib, alectinib) and/or lorlatinib
  * Cohort 2: Prior 1st generation ALK TKI (crizotinib) and/or prior 2nd generation TKI (ceritinib, brigatinib, alectinib) and/or lorlatinib, and platinum-doublet chemotherapy
  * Cohort 3: Prior 1st generation ALK TK (crizotinib) and/or prior 2nd generation TKI (ceritinib, brigatinib, alectinib) and/or lorlatinib, platinum-doublet chemotherapy, and any other number of antineoplastic agents (including immunotherapy, standard or investigational)
* Age ≥ 18
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Absolute neutrophil count (ANC) ≥ 1500/mcL
* Platelets ≥ 100,000/mcL
* Hemoglobin ≥ 9 g/dL without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment)
* Measured or calculated creatinine clearance (CrCl) ≥ 50mL/min (calculated per Cockcroft-Gault formula)
* Serum total bilirubin ≤ 1.5 X upper limit of normal (ULN) (per institutional guidelines) OR direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases
* Alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases
* Albumin ≥ 2.5g/dL
* Female subject of childbearing potential should have a negative serum pregnancy test within 21 days of enrollment prior to receiving the first dose of study medication
* Female subjects of childbearing potential must be willing to use a highly effective method of contraception for the course of the study, through 180 days after the last dose of study medication. Note: Abstinence is acceptable, if patient documents that this is their usual lifestyle or preferred contraception method
* Male subjects of childbearing potential must agree to use an adequate method of contraception starting with the first dose of study therapy through 4 months after the last dose of study therapy. Note: Abstinence is acceptable, if patient documents that this is their usual lifestyle or preferred contraception method
* Ability to swallow pills orally and per investigator's assessment, do not have any significant issues limiting absorption of drug
* Ability to understand and the willingness to sign a written informed consent
* Measurable disease per RECIST v1.1 criteria assessed per screening imaging
* If a cancerous lesion is easily and safely accessible, a pre-treatment biopsy of this lesion is strongly encouraged but NOT required prior to first dose of gilteritinib. Archival or fresh tissue biopsy may be used as long as it was obtained prior to cycle 1 day 1 (C1D1)
* At least 7 days must have elapsed since last anti-neoplastic TKI, chemotherapy, immunotherapy, or investigational agent prior to the first dose of gilteritinib

Exclusion Criteria:

* Received palliative radiation within 7 days of enrollment
* Received prior therapy with a FLT3 inhibitor
* Has a concurrent active malignancy receiving interventional therapy unless it is the investigator's opinion that the concurrent active malignancy will NOT significantly impact the survival of the patient (i.e. early stage breast cancer or prostate cancer on hormonal therapy, basal cell carcinoma awaiting Moh's or other surgery and the respective interventional therapy does NOT interact or interfere with gilteritinib.
* Has known active and symptomatic central nervous system (CNS) metastases and/or carcinomatous meningitis.

  * Subjects with previously treated brain metastases may participate provided they are stable (clinically asymptomatic, and ≥ 2 weeks since completion of treatment) and are not using steroids for at least 7 days prior to enrollment. A repeat MRI brain is not necessary to document stability
  * Patients with carcinomatous meningitis are excluded regardless of clinical stability
* If a patient is found to have new/enlarging brain metastases on the screening MRI, the patient may be monitored closely and radiation could be delayed if the patient has no symptoms, there is no vasogenic edema, and there is no evidence of midline shift.

  * If the patient is symptomatic, there is vasogenic edema, and/or there is midline shift, the patient will need to undergo treatment for these brain metastases and meet exclusion criteria #4 exception to treated brain metastases prior to enrollment. A new MRI brain is NOT required in this situation
* Is pregnant, breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with informed consent through 180 days after the last dose of trial treatment
* Has Child-Pugh class C cirrhosis from any cause
* Mean triplicate screening electrocardiogram (EKG) corrected QT (QTc) > 480 ms
* Grade 3 or 4 NYHA (New York Heart Association) congestive heart failure, unless screening echocardiogram obtained prior to enrollment showed a LVEF (left ventricular ejection fraction) ≥ 45%
* Surgery within 4 weeks prior to first study dose
* Requires treatment with concomitant drugs that are strong inducers of cytochrome P450 (CYP)3A
* Requires treatment with concomitant drugs that are strong inhibitors or inducers of P-glycoprotein (P-gp) with the exception of drugs that are considered absolutely essential for the care of the patient
* Requires treatment with concomitant drugs that target serotonin 5-hydroxytryptamine receptor 1 (5HT1R) or 5-hydroxytryptamine receptor 2B (5HT2BR) or sigma nonspecific receptor, with the exception of drugs that are considered absolutely essential for the care of the patient
* Active/untreated hepatitis B virus (HBV) or hepatitis C virus (HCV) infection; patients with treated HBV and HCV are allowed as long as they meet the AST/ALT and bilirubin criteria
* Known hypersensitivity to gilteritinib or any of the excipients
* Active and clinically significant pancreatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 30 days after last dose of gilteritinib
  Safety will be assessed by the Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0.
Dose-limiting toxicities (DLT) | Cycle 1 day 1 up to cycle 2 day 1 (each cycle is 21 days)
  Toxicities will be assessed by CTCAE v 5.0. DLT's will be defined as >= grade 4 hematologic toxicities, >= grade 3 febrile neutropenia, >= grade 3 non-hematologic toxicities, and posterior reversible encephalopathy syndrome of any grade. Toxicity will be quantified by reporting the proportion of patients who experience a DLT at the identified maximum tolerated dose and by reporting a 95% confidence interval for this proportion.

SECONDARY OUTCOMES:
Anti-tumor response | Up to 2 years after last dose of gilteritinib
  Will be assessed by Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1. Best responses including complete response, partial response, stable disease and progressive disease will be determined by independent radiology assessment.
Progression-free survival (PFS) | From start of treatment to time of progression, assessed up to 2 years after last dose of gilteritinib
  Determined by RECIST v 1.1.
Overall survival (OS) | Cycle 1 day 1 of study start to date of death from any cause, assessed up to 2 years from last dose of gilteritinib
  Median OS and associated 95% confidence intervals will be assessed and reported using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Angel Qin, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (3):
- United States (3):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Georgetown University, Washington D.C., District of Columbia
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No